CLINICAL TRIAL: NCT06361784
Title: "Improving the Success Rate for Thoracic Radiotherapy Through Specific Cardiac Substructure Dosimetry: Location Matters - a Prospective Study"
Brief Title: Improving the Success Rate for Thoracic Radiotherapy Through Specific Cardiac Substructure Dosimetry: Location Matters. (LOCATION MATTERS)
Acronym: LM
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Sponsor
Other Study IDs: INT216-23; MFAG27480 (Other Grant/Funding Number: AIRC Foundation for Cancer Research in Italy)
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-11

CONDITIONS: Locally Advanced Lung Non-Small Cell Carcinoma
Keywords: cardiotoxicity; adverse events; heart substructures; MACE; subclinical warnings
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prospective study LOCATION MATTERS aims to investigate the radiation-induced damage to the heart and the cardiovascular system in patients treated with thoracic radiotherapy. Patients enrolled in the study will complete a set of extensive measures at the baseline, end of RT, and 9 months after treatment. Ultrasound exams, CT scans, pulmonary tests and wearable devices will assess functional and morphological parameters and the association with their variation and the dose delivered to the heart substructures and to the normal lung.

DETAILED DESCRIPTION:
A cohort of locally advanced lung cancer patients treated with RT will be enrolled at Fondazione IRCCS Istituto dei Tumori. Comorbidities and cardiovascular risk factors will be recorded for all the patients. Heart substructures will be automatically contoured on each patient to provide details on the dose distribution.

The investigators will plan an extensive set of cardiac tests before, at the end of RT and 8 months after treatment (to assess cardiac remodelling and pt recovery). It will include an electrocardiogram, echo cardio, spirometry, blood circulating biomarkers (Troponin and Natriuretic peptide tests) and cardiac calcium score from CT. In addition, the researchers will include a set of measures by the use of a vascular ultrasound machine. This machine will allow the investigation of subclinical vascular organ damage indicators, including carotid distention and intima-media thickness (descriptor of the carotid inflammatory state), through a simultaneous and automatic procedure from raw imaging data. This guarantees the extraction of highly reproducible and operator-independent features. Finally, the project will provide smartwatch devices to the patients aiming to get longitudinal information on heart rate, breathe per minute, stress level, Pulse Ox and recovery time after customised exercises.

The study's aim is to associate the most "radiosensitive" functional parameters or biomarkers (i.e. the more prone to vary after RT) with the dose delivered to the HSs. First, researchers will analyze the variations of the parameters in patients with doses above and below the identified constraints from the literature. Second, investigators will test whether a dose relationship model can continuously describe the changes for the parameters with statistically significant differences. The primary focus will be the comprehension of the dose response for morphological and functional parameters that are altered chronically, i.e. with more compromised values at the 1-year measurement.

For this study, the investigators estimate to enrol 150 lung cancer patients in 3 years.

Information on the OS and MACEs will be registered during the clinical standard FU.

Researchers expect to fulfil an FU rate of 90% two years after RT completion. Registering MACEs during the FU time will allow to perform a first direct comparison of the competing part of Task 1.3.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSCLC
* Patients with locally advanced disease (Stage 3)
* Patients treated with RT at Fondazione IRCCS Istituto Nazionale dei Tumori

Exclusion Criteria:

* Previous thoracic radiotherapy
* Previous heart surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include consecutive NSCLC patients with locally advanced disease treated with RT at Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2029-03-29 (Estimated); Study Completion 2029-03-29 (Estimated)

PRIMARY OUTCOMES:
Variation in eco-cardio and eco-vascular parameters after thoracic radiotherapy | Baseline - End RT - 9 months after RT completion
  A set of ultrasound parameters will be normalised to the individual patient value at the baseline. We will evaluate an acute reaction (end of RT) and a late reaction/recovery assessment at 9 months after RT

SECONDARY OUTCOMES:
Major adverse cardiac events post-RT | Baseline - End RT - 9 months after RT completion
  MACEs will be evaluated and recorded during patient FU as a no/yes variable
Increase in cardiac calcification after RT | Baseline - End RT - 9 months after RT completion
  Calcification will be assessed through automatic software able to detect calcifications in the heart based on CT scans. Values will be compared with the baseline

OTHER OUTCOMES:
Longitudinal variation of cardiopulmonary functional parameters | Daily evaluations from baseline to 9 months of FU
  A set of parameters will be assessed through the use of a smartwatch device. Variation with time will be compared to identify risk factors associated to patterns in time evolution.
Texture variation in the heart substructures | Baseline - End RT - 9 months after RT completion
  Quantitative image analysis will be performed on protocol CT scans to assess morphology and tissue composition

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided